CLINICAL TRIAL: NCT06930586
Title: An Observational Study on the Prognostic Value of Neurometabolic Networks in Colorectal Cancer
Brief Title: Prognostic Value of Neurometabolic Networks in CRC (PVNM-CRC)
Acronym: PVNM-CRC
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, yujie bai, MD, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: ybai; 2024M752975 (Other Grant/Funding Number: the China Postdoctoral Science Foundation)
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Brain Injury
MeSH Terms: conditions — Neoplasms; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Cancer: 1. Entry Criteria Male/Female subjects with rectal cancer of at least 18 years of age will be enrolled in this trial.
  2. Subject Inclusion Criteria
  In order to be eligible for participation in this trial, the subject must:
  1. Be ≥ 18 years of age on day of enrollment.
  2. Have pathologically confirmed as rectal adenocarcinoma by electronic colonoscopy biopsy.
  3. Have been diagnosed as colorectal cancer (CRC) by enhanced PET/CT.
  4. Images of PET/CT sequences are available.
  5. Be willing and able to provide written informed assent for Collection and Application of Clinical Sample and Medical Data certified and approved by local ethics committee. Requirements of informed consent for the trial is waived.
  6. . Demonstrate adequate organ function as defined.

SUMMARY:
Colorectal cancer (CRC), with annually increasing incidence and mortality worldwide, has become the second leading cause of cancer-related death. The development of CRC often follows the canonical normal-adenoma-carcinoma (N-A-C) sequence driven by progressive accumulation of molecular genetic events, highlighting the importance of early detection and removal of precancerous lesions. However, some patients who have had adenomas removed still have a high risk of developing new adenomas or CRC, especially for those with chronic or systemic disease, indicating that a compositive regulatory network is involved in the tumorigenesis of CRC. Additionally, despite advances in therapeutic strategies having improved the prognosis of CRC patients, tumor metastasis continues to be the predominant cause of mortality. These suggest the need to transcend limitations focusing solely on intertumoral microenvironment or single-timepoint event but adopt a more systemic perspective to elucidate the mechanisms underlying the whole sequence of CRC development and progression.

The gastrointestinal (GI) tract comprises a complex ecosystem with extensive interactions between normal or neoplastic epithelial cells with immune, neuronal, and other cell types, as well as microorganisms and metabolites within the gut lumen. Specifically, the intricate relationship between the GI tract and the central nervous system (CNS), collectively known as the brain-gut axis, plays a pivotal role in the pathogenesis of gastrointestinal disorders and neoplasm. For instance, chronic stress increased the risk of colon cancer via activating the COX-2/PEG2 system and promoted tumor cell dissemination by remodeling lymph vasculature. The bidirectional communications of the brain-gut axis are generally found to be mediated by neurotransmitters, inflammatory cytokines, metabolites, or gut microbiota. Nonetheless, the spotlight has shone primarily on the brain-gut crosstalk mechanisms in experimental cellular or animal models, with less attention paid to the structural and functional alterations on the brain networks at the patient level.

The evolution of functional neuroimaging modalities and neuroscience technologies has enabled accurate delineation of CNS activities. Specifically, nuclear medicine imaging technology using 2-18F fluoro-2-deoxy-D-glucose (18F-FDG) to adopt whole-body imaging information, is the optimal in vivo method for the investigation of regional human brain metabolism and associations with systemic disorders. We have previously identified the neuronal metabolic-ventricular dyssynchronization axis which might related to major arrhythmic events using myocardial perfusion imaging and the brain 18F-FDG positron emission tomography (PET). Given the potential dual interactions of the brain-gut axis, identification of specific brain regions associated with CRC development and progression might lead to a better understanding of the disease's neurobiological underpinnings and inform the development of targeted therapeutic strategies.

Hence, this study was structured to elucidate the role of neuro-metabolism and its potential mediator in regulating CRC tumorigenesis and metastasis. By delving into the neurometabolic-gut axis in CRC, the resulting mechanistic insights might be leveraged to identify diagnostic and prognostic biomarkers and to develop novel therapeutic interventions for CRC patients.

DETAILED DESCRIPTION:
OBJECTIVE(S) & HYPOTHESIS(ES) Objective: Evaluate area under curve (AUC) of BRIDGE in predicting overall survival (OS) for CRC patients. Compare the AUC of BRIDGE with clinical prediction models in predicting survival status for CRC patients. Evaluate the sensitivity, specificity, positive prediction value (PPV) and negative prediction value (NPV)of BRIDGE in predicting OS for CRC patients.

Hypothesis: BRIDGE achieves an AUC over 0.80 in predicting OS for CRC patients. BRIDGE is superior to clinical prediction models in terms of AUC in predicting OS for CRC patients.

BACKGROUND & RATIONALE Colorectal cancer (CRC), with annually increasing incidence and mortality worldwide, has become the second leading cause of cancer-related death. The gastrointestinal (GI) tract comprises a complex ecosystem with extensive interactions between normal or neoplastic epithelial cells with immune, neuronal, and other cell types, as well as microorganisms and metabolites within the gut lumen. Specifically, the intricate relationship between the GI tract and the central nervous system (CNS), collectively known as the brain-gut axis, plays a pivotal role in the pathogenesis of gastrointestinal disorders and neoplasm. For instance, chronic stress increased the risk of colon cancer via activating the COX-2/PEG2 system and promoted tumor cell dissemination by remodeling lymph vasculature. The bidirectional communications of the brain-gut axis are generally found to be mediated by neurotransmitters, inflammatory cytokines, metabolites, or gut microbiota. Nonetheless, the spotlight has shone primarily on the brain-gut crosstalk mechanisms in experimental cellular or animal models, with less attention paid to the structural and functional alterations on the brain networks at the patient level.

The evolution of functional neuroimaging modalities and neuroscience technologies has enabled accurate delineation of CNS activities. Specifically, nuclear medicine imaging technology using 2-18F fluoro-2-deoxy-D-glucose (18F-FDG) to adopt whole-body imaging information, is the optimal in vivo method for the investigation of regional human brain metabolism and associations with systemic disorders. The investigators have previously identified the neuronal metabolic-ventricular dyssynchronization axis which might related to major arrhythmic events using myocardial perfusion imaging and the brain 18F-FDG positron emission tomography (PET). Given the potential dual interactions of the brain-gut axis, identification of specific brain regions associated with CRC development and progression might lead to a better understanding of the disease's neurobiological underpinnings and inform the development of targeted therapeutic strategies. Hence, this study was structured to elucidate the role of neuro-metabolism and its potential mediator in regulating CRC tumorigenesis and metastasis. By delving into the neurometabolic-gut axis in CRC, the resulting mechanistic insights might be leveraged to identify diagnostic and prognostic biomarkers and to develop novel therapeutic interventions for CRC patients.

Previously, investigators have constructed a BRIDGE based on retrospective datasets. The study is conducted to further prospectively verify the clinical applicability and generalizability of BRIDGE in predicting OS for CRC patients. The prediction performance of BRIDGE will be evaluated in a prospective dataset, and compared to conventional clinical-based prediction models in the trial, which might potentially provide important evidence for the feasibility and clinical value of integration of brain images for artificial intelligence-aided GI cancer medicine.

The primary accuracy endpoint in the study is the AUC, a significant indicator of classification performance of a binary classifier, which has been widely used to evaluate model performance in the field of machine learning.

METHODOLOGY Inclusion Criteria

1. Age ≥ 18 years. 2. Have pathologically confirmed as colorectal adenocarcinoma. 3. Have been diagnosed as colorectal cancer (CRC) by PET/CT. 4. Images of PET/CT sequences are available. Exclusion Criteria

1. Has a concomitant additional malignancy that is processing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
2. Have a history of cerebrovascular disease (CVD), refers to a general term for a class of diseases in which cerebrovascular lesions lead to brain dysfunction, including cerebrovascular stenosis, brain localized or diffuse brain dysfunction caused by various cerebrovascular lesions such as vascular occlusion, cerebrovascular rupture, cerebrovascular malformations, or cerebrovascular injuries in doctoral dissertations of Capital Medical University, mainly including ischemic stroke and hemorrhagic stroke, defined as cerebrovascular diseases caused by organic brain injury with sudden onset, rapid onset of localized or diffuse brain function defects as clinical features.

   Have a major neuropsychiatric abnormality, or had a life expectancy of fewer than 3 months.
3. Have a history of mental illness, including but not limited to parkinsonism, depression, anxiety, schizophrenia, or dementia.
4. Have a history of severe head trauma.
5. Have a history or current evidence of any condition, laboratory abnormality, or substance abuse disorders that might confound the results of trial or interfere with the subject's participation for the full duration of the trial.
6. Have a history of acute cardiovascular events within 4 weeks before enrollment, including but not limited to acute coronary syndrome, acute decompensated heart failure, and malignant arrhythmia; have a non-tumor condition limiting life expectancy to less than 1 year.
7. Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
8. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to treatment initiation.
9. Have an active infection requiring systemic therapy.
10. Be pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial.
11. Lack of images of PET/CT, or insufficient quality of PET/CT images to obtain measurements.
12. Be currently participating in an additional trial and receiving study therapy. Subject Withdrawal/Discontinuation Criteria The subject discontinues/withdraws study during the trial. Basic Information Collection and Serial Number Generation Once enrollment, the basic information including demographics and baseline clinical characteristics of each subject will be recorded. A unique tracking number will be generated randomly for each subject that will be used to identify the subject for all procedures in the trial.

Imaging Data Collection and Process PET/CT Imaging Collection and Anonymization For each subject, initial tumor imaging by PET/CT should have been performed within 1-2 weeks after enrolled. The process for imaging collection and transmission is manipulated in a uniform imaging protocol by radiologists and technicians in participating institutions. The whole series of PET/CT scans should be exported as DICOM files and completely anonymized with unique tracking number before uploaded to the designated cloud platform.

PET/CT Imaging Quality Control Images of PET/CT scans acquired in sites will be downloaded and reviewed by an independent radiologist experienced in PET/CT in the central laboratory to ensure high image quality

ELIGIBILITY:
Male/Female subjects with rectal cancer of at least 18 years of age will be enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Entry Criteria Male/Female subjects with rectal cancer of at least 18 years of age will be enrolled in this trial.
  2. Subject Inclusion Criteria
  In order to be eligible for participation in this trial, the subject must:
  2.1. Be ≥ 18 years of age on day of enrollment. 2.2. Have pathologically confirmed as rectal adenocarcinoma by electronic colonoscopy biopsy.
  2.3. Have been diagnosed as colorectal cancer (CRC) by enhanced PET/CT. 2.4. Images of PET/CT sequences are available. 2.5. Be willing and able to provide written informed assent for Collection and Application of Clinical Sample and Medical Data certified and approved by local ethics committee. Requirements of informed consent for the trial is waived.
  2.6.. Demonstrate adequate organ function as defined in Table 1. All screening labs should be performed within 10 days of treatment initiation.
Sampling Method: Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) | From March 1, 2024 to December 31, 2026-31
  AUC is defined as the probability that a randomly chosen positive example is ranked higher than a randomly chosen negative example. A higher AUC indicates a better classification performance of a definite predictor. The AUC is evaluated by calculating the area under curve of receiver operating characteristics (ROC) which plots the proportion of true positive cases (sensitivity) against the proportion of false positive cases (1-specificity) based on various predictive probability threshold. The 95% confidence intervals (95%CI) of AUC are generated by bootstrapping strategy in 1000 sampling times.

CONTACTS AND LOCATIONS:
Locations (1):
- PET/CT, Henan, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
CONFIDENTIALITY AND DATA SHARING PLAN
  1. Confidentiality of Data Data generated in the trials will be considered confidential by the investigators, except to the extent that it is included in a publication. During the trial, the subject will be identified by unique tracking number.
  2. Data Sharing Plan The subject data (deidentified participant information and PET/CT data) and the full study protocol will be made available to the scientific community, immediately on publication, with as few restrictions as possible. All requests should be submitted to the investigators for consideration. A data use agreement will be required before the release of subject data and institutional review board approval as appropriate.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From December 31, 2027 to December 31, 2030-31
Access Criteria: The subject data (deidentified participant information and PET/CT data) and the full study protocol will be made available to the scientific community, immediately on publication, with as few restrictions as possible. All requests should be submitted to the investigators for consideration. A data use agreement will be required before the release of subject data and institutional review board approval as appropriate.

REFERENCES:
- [Background] Schledwitz A, Xie G, Raufman JP. Exploiting unique features of the gut-brain interface to combat gastrointestinal cancer. J Clin Invest. 2021 May 17;131(10):e143776. doi: 10.1172/JCI143776. PMID 33998603
- [Background] Leslie A, Carey FA, Pratt NR, Steele RJ. The colorectal adenoma-carcinoma sequence. Br J Surg. 2002 Jul;89(7):845-60. doi: 10.1046/j.1365-2168.2002.02120.x. PMID 12081733
- [Background] Murphy CC, Zaki TA. Changing epidemiology of colorectal cancer - birth cohort effects and emerging risk factors. Nat Rev Gastroenterol Hepatol. 2024 Jan;21(1):25-34. doi: 10.1038/s41575-023-00841-9. Epub 2023 Sep 18. PMID 37723270
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- See also: Related Info — https://github.com/StandWisdom/Radiopathomics-pCR-nCRT